CLINICAL TRIAL: NCT02967679
Title: SERENDEM Study: MD1003 in Patients Suffering From Demyelinating Neuropathies, an Open Label Pilot Study
Brief Title: SERENDEM : MD1003 in Patients Suffering From Demyelinating Neuropathies, an Open Label Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedDay Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MD1003CT2015-01 SERENDEM
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Peripheral Neuropathy; Charcot-Marie-Tooth Disease; Charcot-Marie-Tooth Disease Type 1A; Charcot-Marie-Tooth Disease, Type 1B; Anti-MAG Neuropathy
Keywords: Neuropathy; Demyelinating polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Peripheral Nervous System Diseases; Charcot-Marie-Tooth Disease | interventions — Biotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MD1003 (Experimental): MD1003 100mg capsules, 1 capsule tid for 48 weeks
  Interventions: Drug: MD1003

INTERVENTIONS:
Drug: MD1003
  Other Names: High Dose Biotin

SUMMARY:
The single-center, open-label Phase II study has the objective of assess the effect of MD1003 on motor and sensory conduction in patients suffering from demyelinating polyneuropathies in 15 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged between 20 and 85 years.
* Patients fulfilling one of the following diagnosis:
* Five patients with chronic inflammatory demyelinating polyneuropathy on both clinical and neurophysiological grounds.
* Five patients with proven genetic diagnosis of CMT1a or CMT1b
* Five patients with anti-MAG polyneuropathy.
* Electrophysiological parameters worsening for the past 3 years
* Available EMG record, performed during the past 6 months to assess variability of NCV parameters
* Signed and dated written informed consent to participate in the study in accordance with local regulations
* Likely to be able to participate in all scheduled evaluation and complete all required study procedures,
* In the opinion of the investigator, the patient will be compliant and have a high probability of completing the study.
* Both male and female subjects who are not either surgically sterile (tubal ligation/obstruction or removal of ovaries or uterus) or post-menopausal (no spontaneous menstrual periods for at least one year confirmed by a negative hormone panel) must commit to using TWO highly effective method of birth control for the duration of the study and for two months after the treatment termination.

Exclusion Criteria:

* Any general chronic handicapping disease other than peripheral neuropathy
* Impossibility to perform the 10 meters walking test
* Impossibility to assess electrophysiological parameters
* Patients with uncontrolled hepatic disorder, renal or cardiovascular disease, or cancer,
* Patients with hypersensitivity to MD1003 excipients (lactose)
* Laboratory tests out of normal range according to the reference laboratory values. Deviations may be accepted if considered by the investigator as not clinically significant with regards to the study continuation,
* Patients with history or presence of alcohol abuse or drug addiction,
* Patients likely to be non-compliant to the study procedures or for whom a long-term follow-up seems to be difficult to achieve.
* Any new medication for neuropathy initiated less than 3 months prior to inclusion. For CIDP patients, relapse in the past 3 months before inclusion.
* Not easily contactable by the investigator in case of emergency or not capable to call the investigator
* Subjects without effective contraception

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain CREANGE, MD, Principal Investigator — Hôpital Henri Mondor, Créteil, France; Frederic Sedel, MD, Study Director — Medday Pharmaceuticals
Locations (1):
- Hôpital Henri Mondor, Créteil, France, Créteil, France

REFERENCES:
- [Derived] Creange A, Hutin E, Sedel F, Le Vigouroux L, Lefaucheur JP. High-dose pharmaceutical-grade biotin in patients with demyelinating neuropathies: a phase 2b open label, uncontrolled, pilot study. BMC Neurol. 2023 Oct 30;23(1):389. doi: 10.1186/s12883-023-03440-y. PMID 37899433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MD1003
Started | 15
Completed | 14
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: * Five patients with chronic inflammatory demyelinating polyneuropathy on both clinical and neurophysiological grounds.
  * Five patients with proven genetic diagnosis of CMT1a or CMT1b
  * Five patients with anti-MAG polyneuropathy.
Arm/Group | MD1003
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.36 (14.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 15
Disease type [Number; unit: participants]
  CIDP patients | 5
  CMT1a or CMT1b patients | 5
  anti-MAG polyneuropathy | 5

OUTCOME MEASURES:

1. Primary Outcome: Motor Nerve Conduction Velocity (m/Sec)
Description: Absolute change from baseline at Week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | MD1003
Number analyzed (Participants) | 15
m/s | 1.67 (11.45)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.7615, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.67, Standard Deviation 11.45

2. Primary Outcome: Distal Latency (Msec)
Description: Absolute change from baseline at Week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | MD1003
Number analyzed (Participants) | 15
ms | 0.20 (8.89)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.5995, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.20, Standard Deviation 8.89

3. Primary Outcome: F Wave Latency (Msec)
Description: Absolute change from baseline at Week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | MD1003
Number analyzed (Participants) | 9
ms | 4.8 (8.40)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.1641, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 4.8, Standard Deviation 8.40

4. Primary Outcome: Length of Motor Nerve Potential
Description: Absolute change from baseline at W48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | MD1003
Number analyzed (Participants) | 15
ms | 8.5 (16.50)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.0353, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 8.5, Standard Deviation 16.5

5. Secondary Outcome: ONLS (Overall Neuropathy Limitations Scale)
Description: The ONLS focuses on upper and lower limb functions, and consists of a checklist for interviewing patients. It is scored from 0 to 5 on the upper limb section and from 0 to 7 on the lower limb section. A score of 0 indicates no limitations (the ceiling of the scale) and a score of 5 or 7 indicates no purposeful movement. Absolute change from baseline at week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MD1003
Number analyzed (Participants) | 15
score on a scale | -0.5 (1.4)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.2642, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.5, Standard Deviation 1.4

6. Secondary Outcome: Change From Baseline at Week 48 for Timed 10-meter Walk Test
Description: Absolute change from baseline at week 48. The patient is instructed to walk at normal pace for 10 meters. Start and stop of performance time coincides with the toes of the leading foot crossing the 2-m mark and the 8-m mark, respectively. From these data, the speed may be calculated by dividing the middle 6 m by the time (in seconds).
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: second
Arm/Group | MD1003
Number analyzed (Participants) | 15
second | -0.6 (1.2)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.1777, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -0.6, Standard Deviation 1.2

7. Secondary Outcome: Absolute Change From Baseline at Week 48 for Medical Research Council (MRC) Subscore (Total Muscle) and Total Score
Description: MRC score assessed in 19 muscles.
  The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
  The patient's effort is graded on a scale of 0-5:
  Grade 5: Muscle contracts normally against full resistance. Grade 4: Muscle strength is reduced but muscle contraction can still move joint against resistance.
  Grade 3: Muscle strength is further reduced such that the joint can be moved only against gravity with the examiner's resistance completely removed. As an example, the elbow can be moved from full extension to full flexion starting with the arm hanging down at the side.
  Grade 2: Muscle can move only if the resistance of gravity is removed. As an example, the elbow can be fully flexed only if the arm is maintained in a horizontal plane.
  Grade 1: Only a trace or flicker of movement is seen or felt in the muscle or fasciculations are observed in the muscle.
  Grade 0: No movement is observed.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MD1003
Number analyzed (Participants) | 15
score on a scale | 4.5 (8.2)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.0371, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 4.5, Standard Deviation 8.2

8. Secondary Outcome: INCAT Sensory Sum Score (ISS)
Description: This sensory scale comprises pin prick and vibration sense plus a two point discrimination value in the arms and legs, and ranges from 0 ("normal sensation") to 20 ("most severe sensory deficit"). Absolute change from baseline at week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MD1003
Number analyzed (Participants) | 15
score on a scale | -2.2 (2.9)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.0142, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -2.2, Standard Deviation 2.9

9. Secondary Outcome: 6-minute Walk Test
Description: The 6MWT is a practical simple test that requires a 30 m (100-ft) hallway. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. Absolute change from baseline at week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: m
Arm/Group | MD1003
Number analyzed (Participants) | 15
m | 61.1 (48.9)

10. Secondary Outcome: Posturography Score
Description: Computerized dynamic posturography (CDP) is a non-invasive specialized clinical assessment technique used to quantify the central nervous system adaptive mechanisms (sensory, motor and central) involved in the control of posture and balance, both in normal and abnormal conditions. Absolute change of speed in spontaneous speed condition from baseline at week 48.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | MD1003
Number analyzed (Participants) | 13
m/s | 0.111 (0.201)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.1055, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.111, Standard Deviation 0.201

11. Secondary Outcome: Excitability Testing: Supernormality (%)
Description: Nerve excitability testing is a non-invasive approach in investigating the pathophysiology of peripheral nerve disorders, which determines the electrical properties of the nerve membrane at the site of stimulation. Absolute change from baseline at week 48.
  After a nerve fiber is depolarized, a sequence of excitability changes, called the 'recovery cycle', occurs before the membrane potential returns to its resting stage. This cycle includes phases in which the nerve excitability is decreased ('refractory period' or increased ('supernormal period'). During the 10-30 ms following the end of the refractory period, the axon increases its excitability and the nerve fiber is more easily excited (the supernormal period). Depolarization of the node of Ranvier excites the adjacent internodes, which then charge with electric current as capacitors. Supernormality depends on many factors and its interpretation is therefore not univoqual. Data were provided for information only.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of supernormality
Arm/Group | MD1003
Number analyzed (Participants) | 15
percentage of supernormality | 9.84 (28.16)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.2130, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 9.84, Standard Deviation 28.16

12. Secondary Outcome: Strength-duration Time Constant (ms)
Description: This secondary outcome measure is an electrophysiological testing endpoint. Absolute change from baseline at week 48.
  Strength-duration Time Constant (ms) is a measurement of excitability, defined as the duration of the stimulus that has twice the strength of the rheobase current (see below). The lower the rheobase is, the higher is the Strenght duration time constant. Accordingly, higer values of SDTC are associated with better outcome.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | MD1003
Number analyzed (Participants) | 15
ms | 0.068 (0.112)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.0393, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.068, Standard Deviation 0.112

13. Secondary Outcome: Rheobase (mA)
Description: This secondary outcome measure is an electrophysiological testing endpoint. Absolute change from baseline at week 48.
  Rheobase is the minimal strength of an electrical stimulus of infinitely long duration that is able to cause excitation. Low values are associated with better outcome (the nerve becomes more excitable).
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | MD1003
Number analyzed (Participants) | 15
mA | -5.905 (6.283)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.0004, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -5.905, Standard Deviation 6.283

14. Secondary Outcome: Refractoriness (%)
Description: This secondary outcome measure is an electrophysiological testing endpoint. Absolute change from baseline to week 48.
  After a nerve fiber is depolarized, a sequence of excitability changes, called the 'recovery cycle', occurs before the membrane potential returns to its resting stage. This cycle includes phases in which the nerve excitability is decreased ('refractory period' or increased ('supernormal period'). Refractoriness depends on many factors and its interpretation is therefore not univoqual. Data were provided for information only.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: percentage of refractoriness
Arm/Group | MD1003
Number analyzed (Participants) | 15
percentage of refractoriness | -4.28 (32.21)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.3303, Wilcoxon (Mann-Whitney); Mean Difference (Net) = -4.28, Standard Deviation 32.21

15. Secondary Outcome: Minimum Absolute Refractory Period (ms).
Description: This secondary outcome measure is an electrophysiological testing endpoint. Absolute change from baseline at week 48.
  After a nerve fiber is depolarized, a sequence of excitability changes, called the 'recovery cycle', occurs before the membrane potential returns to its resting stage. This cycle includes phases in which the nerve excitability is decreased ('refractory period' or increased ('supernormal period'). Refractoriness depends on many factors and its interpretation is therefore not univoqual. Data were provided for information only.
Time Frame: 48 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | MD1003
Number analyzed (Participants) | 15
ms | 0.000 (0.092)
Statistical Analysis 1: Comparison: MD1003; Test type: Other; p = 0.9229, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.000, Standard Deviation 0.092

16. Secondary Outcome: Maximum Absolute Refractory Period (ms).
Description: as for outcome 15
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | MD1003
Number analyzed (Participants) | 15
ms | -0.277 (0.871)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | MD1003
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MD1003 (N=15)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Autoimmune encephalopathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MD1003 (N=15)
Insomnia (Nervous system disorders) | 3 (3)
Gastric disorder (Gastrointestinal disorders) | 1 (1)
balance disorder (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (2)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Burn oesophageal (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Laboratory test interference (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Breast reconstruction (Surgical and medical procedures) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT02967679/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT02967679/SAP_001.pdf